CLINICAL TRIAL: NCT06197308
Title: Evaluation of an Oral Microbiota-based Therapeutic as a Treatment Option for Primary Sclerosing Cholangitis
Brief Title: Evaluation of an Oral Microbiota-based Therapeutic as a Treatment Option for PSC
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-2023-32551
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Vancomycin; Amoxicillin

STUDY DESIGN:
Intervention Model Description: Adult patients with PSC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PCS patients (Experimental)
  Interventions: Drug: oral vancomycin and oral amoxicillin

INTERVENTIONS:
Drug: oral vancomycin and oral amoxicillin — In this study, PSC patients will receive an antibiotic preconditioning regimen of oral vancomycin (500 mg liquid twice a day) for 28 days and oral amoxicillin (1000 mg twice a day) for 7 days (during the last 7 days of the oral vancomycin). Following vancomycin and amoxicillin, encapsulated, freeze-dried microbiota preparation (MTP-101C) will be administered - dosed at ≥ 5 x 10^11 bacteria (five capsules) daily for 3 days followed by ≥ 2 x 10^11 bacteria (two capsules) for 11 days - for a total of 14 days of MTP-101C; total of 37 capsules.

SUMMARY:
This pilot clinical trial will evaluate the initial safety and feasibility of microbiota transplant therapy (MTT) inpatients with primary sclerosing cholangitis (PSC). This trial will inform development of future trials in treatment of PSC.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-76
* Serum total bilirubin at screening ≤ 2x the upper limit of normal
* Absence of biliary obstruction and malignancy by ultrasound or equivalent imaging within 6 months of study entry
* Anticipated maintenance of current medication regimen through the treatment period (UDCA, azathioprine, corticosteroid, methotrexate, 5-ASA, biologic therapy and/or probiotic)
* 3-month washout period of obeticholic acid or other experimental therapies for PSC
* Stated willingness to comply with all study procedures and availability for the duration of trial to follow-up by telephone, in-person, email, and/or video visits or correspondence.
* Informed consent

Exclusion Criteria:

* Antibiotic therapy (except vancomycin) within 3 months or anticipated antibiotic use in the course of the MTT treatment
* Presence of complications of advanced PSC, such as hepatic encephalopathy, ascites, history of esophageal varices, portal hypertension, hepato-renal syndrome, portopulmonary syndrome, and hepato-pulmonary syndrome
* Evidence for viral hepatitis (history of Hepatitis C is eligible with undetectable HCV RNA); HIV/AIDS
* Metabolic or inherited liver disease (e.g., Wilson's, hemochromatosis, alpha-1-antitrypsin deficiency)
* Another disease involving bile ducts (e.g., primary biliary cholangitis, IgG4-related cholangitis, secondary sclerosing cholangitis)
* Evidence of cirrhosis on the last magnetic resonance cholangiopancreatography (within 6 months)
* Pregnancy or attempting to become pregnant or breastfeeding.
* History of liver transplantation, anticipated need for liver transplantation within 12- months from randomization, or a Model of End Stage Liver Disease (MELD) score of ≥15
* Active malignancy
* Active alcohol overuse (>4 drinks per day for men, and >2 drinks per day for women)
* Moderate-to-severe renal impairment with a calculated creatinine clearance of < 45 mL/min
* Neutropenia (an absolute neutrophil count < 0.5 x 109 cells/L)
* History of allergic reaction to vancomycin
* History of allergic reaction to amoxicillin or other beta-lactam antibiotics
* Any other conditions or abnormalities that, in the opinion of the investigator, may compromise the safety of the subject or interfere with the subject participating in or completing the study
* Total colectomy

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate safety of MTT in patients with PSC | 221 days
  Determine the frequency of serious adverse events and other adverse events
To evaluate feasibility of MTT in patients with PSC | 221 days
  Determine proportion of subjects taking 100% of the MTT per protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Aby, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States